CLINICAL TRIAL: NCT02704143
Title: Stereotactic Body Radiation Therapy With Sequential S-1 for Patients With Locally Advanced Pancreatic Cancer and Poor Medical Conditions --a Phase II Clinical Trial
Brief Title: Combination of SBRT With Sequential S-1 for Treating Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director of Radiation Oncology Department, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Changhai Hosp
Record Dates: First submitted 2016-03-01; First posted 2016-03-09 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Cancer
Keywords: stereotactic body radiation therapy; S-1; locally advanced pancreatic cancer; poor medical conditions
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Intervention Model Description: stereotactic bodt radiation therapy plus sequential S-1 for locally pancreatic cancer
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination of Cyberknife with S-1 (Experimental): Patients with locally advanced pancreatic cancer meeting all inclusion criteria will receive combination of Cyberknife with S-1.
  Interventions: Other: combination of Cyberknife with S-1

INTERVENTIONS:
Other: combination of Cyberknife with S-1 — Radiation therapy combined with chemotherapy

SUMMARY:
The safety and efficacy of combination of SBRT with sequential S-1 in treating patients with locally advanced pancreatic cancer and poor medical conditions will be evaluated.

DETAILED DESCRIPTION:
Although the incidence rate of pancreatic cancer is not as high as that of other gastrointestinal carcinoma in China, the cancer mortalities of males and females ranked the sixth and seventh respectively in 2013, with a surprising low 5-year survival rate (<5%). Only 15%-20% patients are suitable for surgeries among those first diagnosed with pancreatic cancer and the 5-year survival rate of patients with R0 resection is still less than 20%.

Therefore, better efficacy is not available via surgeries alone resulting in great emphasis on adjuvant chemoradiotherapy. In 1997, gemcitabine was confirmed to be the standard chemotherapy for pancreatic cancer. However, it has not been proved that gemcitabine significantly improved prognosis in long term follow-up while some patients are refractory to gemcitabine. Hence, development of more effective chemotherapy is urgent.

S-1 is the prodrug of 5-fluorouracil (5-FU), comprised of tegafur, gimeracil (dihydropyrimidine dehydrogenase inhibitor) and oteracil (the inhibitor of phosphorylation in gastrointestinal tract) with a ratio of 1:0.4:1. The first phase II clinical trials showed good clinical efficacy with S-1.Moreover, Ueno et al. identified better objective response rates with S-1 than those with gemcitabine. Besides, S-1 is not inferior to gemcitabine regarding to overall survival rates and progression free survival rates. And significant improvement of progression free survival rates can be achieved by combination of S-1 and gemcitabine. There was no difference between incidence rates of adverse effects of S-1 and gemcitabine, with more gastrointestinal toxicities with S-1 while more hematologic toxicities with gemcitabine. Therefore, S-1 is an alternative for treating locally advanced or metastatic pancreatic cancer, especially for those resistant to gemcitabine. Although there are no phase III studies on S-1, phase II studies have already shown better disease control rates (52%-58%), median overall survival time (4.5-6.3 months) and tolerable adverse effects in advanced pancreatic cancer resistant to gemcitabine treated with S-1.

Though S-1 is appropriate for advanced pancreatic cancer, it is not superior to gemcitabine with respect to clinical efficacy. In addition, fewer encouraging results are gained with combination of S-1 and other drug. As a result, S-1 combined with radiotherapy is gradually applied in treatment of pancreatic cancer.

5-FU was proved to be radiosensitive thus improving clinical efficacy. S-1 combined with radiotherapy has demonstrated better prognosis with the median overall survival time of 12.9-16.8 months. Furthermore, some patients can be operable after S-1 and radiotherapy.

Compared with conventional radiation, a single-fraction dose and total dose of target volume can be increased in stereotactic body radiation therapy (SBRT). In addition, doses of organs at risk would be reduced, thus effectively improving local control rates and reducing radiation related toxicity. Shorter courses of SBRT also enhance patients' compliance and render the initial of other treatment on schedule possible. Nevertheless, there are few studies focusing on S-1 combined with SBRT for locally advanced pancreatic cancer. Especially for patients with poor medical coonditions, though gemcitabine alone is recommended in the NCCN guideline, S-1 may be a better option due to more adverse effects induced by gemcitabine in Asian. Additionally, local ablative treatment combined with chemotherapy may provide more survival benefits for those patients. Hence, efficacy of combination of S-1 and SBRT needs to be further confirmed. Based on our experience in treating locally advanced pancreatic cancer, SBRT combined with sequential S-1 as the initial treatment for patients with locally advanced pancreatic cancer and poor medical conditions is proposed to evaluate its clinical efficacy.

Study Procedure:

1. CyberKnife SBRT body fixation (vacuum-bag) will be used in immobilizing the body, the arms and the legs. Patients will undergo a plain CT as well as an enhanced pancreatic parenchymal CT for radiation treatment planning and target delineation.
2. SBRT will be delivered on CyberKnife with Synchrony Respiratory Tracking system. The tumor will be tracked with implanted fiducial markers by Fiducial Tracking System. Treatment will be delivered in 5 fractions within 1 to 2 weeks at the discretion of the investigator.
3. A body fixation (vacuum-bag) will be used in immobilizing the body, the arms (both arms are along the body) and the legs.
4. The total doses depend on patients' medical conditions, ranging from 35Gy-40Gy/5Fx.
5. Patients receive 80 mg of S-1 per square meter of body surface area twice a day for 4 weeks, followed by 2 weeks of rest as one course, which would repeat for six cycles.The initiation of S-1 is one month after SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced pancreatic cancer proved by CT or MRI and biopsy
2. Without any other treatment before SBRT
3. A life expectancy of >3months
4. ECOG: 2 or 3 points
5. Age of more than 18 years old
6. Blood routine examination: Absolute neutrophil count (ANC) ≥ 1.5 ×10^9 cells/L, leukocyte count≥ 3.5 ×10^9 cells/L, platelets ≥ 70×10^9 cells/L, hemoglobin ≥ 8.0 g/dl
7. Liver and kidney function tests: Albumin > 2.5 g/dL, total bilirubin < 3 mg/dL, creatinine < 2.0 mg/dL, AST<2.5 × ULN(Upper Limit of Normal)(0-64U/L), ALT<2.5 × ULN(0-64U/L)
8. INR < 2 (0.9-1.1)
9. Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior surgery, chemotherapy or radiation for the pancreatic cancer
2. Evidences of metastatic disease such as nodal or distant metastases by abdomen CT and chest CT or FDG PET-CT
3. Contraindication to receiving radiotherapy
4. ECOG: 0-1 point
5. Age<18
6. Abnormal results of blood routine examinations and liver and kidney tests
7. Patients with active inflammatory bowel diseases or peptic ulcer
8. Gastrointestinal bleeding or perforation within 6 months
9. Heart failure: NYHA III-IV
10. Women who are pregnant
11. Participation in another clinical treatment trial while on study
12. Patients in whom fiducial implantation was not possible
13. Inability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huo Jun Zhang, MD., PH.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Sener SF, Fremgen A, Menck HR, Winchester DP. Pancreatic cancer: a report of treatment and survival trends for 100,313 patients diagnosed from 1985-1995, using the National Cancer Database. J Am Coll Surg. 1999 Jul;189(1):1-7. doi: 10.1016/s1072-7515(99)00075-7. PMID 10401733
- [Background] Richter A, Niedergethmann M, Sturm JW, Lorenz D, Post S, Trede M. Long-term results of partial pancreaticoduodenectomy for ductal adenocarcinoma of the pancreatic head: 25-year experience. World J Surg. 2003 Mar;27(3):324-9. doi: 10.1007/s00268-002-6659-z. Epub 2003 Feb 27. PMID 12607060
- [Background] Tseng JF, Raut CP, Lee JE, Pisters PW, Vauthey JN, Abdalla EK, Gomez HF, Sun CC, Crane CH, Wolff RA, Evans DB. Pancreaticoduodenectomy with vascular resection: margin status and survival duration. J Gastrointest Surg. 2004 Dec;8(8):935-49; discussion 949-50. doi: 10.1016/j.gassur.2004.09.046. PMID 15585381
- [Background] Hoyer M, Roed H, Sengelov L, Traberg A, Ohlhuis L, Pedersen J, Nellemann H, Kiil Berthelsen A, Eberholst F, Engelholm SA, von der Maase H. Phase-II study on stereotactic radiotherapy of locally advanced pancreatic carcinoma. Radiother Oncol. 2005 Jul;76(1):48-53. doi: 10.1016/j.radonc.2004.12.022. PMID 15990186
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Ueno H, Okusaka T, Ikeda M, Takezako Y, Morizane C. An early phase II study of S-1 in patients with metastatic pancreatic cancer. Oncology. 2005;68(2-3):171-8. doi: 10.1159/000086771. Epub 2005 Jul 4. PMID 16006754
- [Background] Ueno H, Ioka T, Ikeda M, Ohkawa S, Yanagimoto H, Boku N, Fukutomi A, Sugimori K, Baba H, Yamao K, Shimamura T, Sho M, Kitano M, Cheng AL, Mizumoto K, Chen JS, Furuse J, Funakoshi A, Hatori T, Yamaguchi T, Egawa S, Sato A, Ohashi Y, Okusaka T, Tanaka M. Randomized phase III study of gemcitabine plus S-1, S-1 alone, or gemcitabine alone in patients with locally advanced and metastatic pancreatic cancer in Japan and Taiwan: GEST study. J Clin Oncol. 2013 May 1;31(13):1640-8. doi: 10.1200/JCO.2012.43.3680. Epub 2013 Apr 1. PMID 23547081
- [Background] Morizane C, Okusaka T, Furuse J, Ishii H, Ueno H, Ikeda M, Nakachi K, Najima M, Ogura T, Suzuki E. A phase II study of S-1 in gemcitabine-refractory metastatic pancreatic cancer. Cancer Chemother Pharmacol. 2009 Jan;63(2):313-9. doi: 10.1007/s00280-008-0741-7. Epub 2008 Apr 9. PMID 18398614
- [Background] Sudo K, Yamaguchi T, Nakamura K, Denda T, Hara T, Ishihara T, Yokosuka O. Phase II study of S-1 in patients with gemcitabine-resistant advanced pancreatic cancer. Cancer Chemother Pharmacol. 2011 Feb;67(2):249-54. doi: 10.1007/s00280-010-1311-3. Epub 2010 Mar 30. PMID 20352216
- [Background] Mizuno N, Yamao K, Komatsu Y, et al. Randomized phase II trial of S-1 versus S-1 plus irinotecan (IRIS) in patients with gemcitabinerefractory pancreatic cancer. J Clin Oncol, 2012, 30 (suppl 34): abstr 263
- [Background] Okusaka T, Ohkawa S, Isayama H, et al. Randomized phase II trial of S-1 versus S-1 plus oxaliplatin (SOX) in patients with GEM refractory pancreatic cancer. ESMO, 2012, abstract 1437
- [Background] Ge F, Xu N, Bai Y, Ba Y, Zhang Y, Li F, Xu H, Jia R, Wang Y, Lin L, Xu J. S-1 as monotherapy or in combination with leucovorin as second-line treatment in gemcitabine-refractory advanced pancreatic cancer: a randomized, open-label, multicenter, phase II study. Oncologist. 2014 Nov;19(11):1133-4. doi: 10.1634/theoncologist.2014-0223. Epub 2014 Oct 1. PMID 25273077
- [Background] Rich TA, Shepard RC, Mosley ST. Four decades of continuing innovation with fluorouracil: current and future approaches to fluorouracil chemoradiation therapy. J Clin Oncol. 2004 Jun 1;22(11):2214-32. doi: 10.1200/JCO.2004.08.009. PMID 15169811
- [Background] Moningi S, Marciscano AE, Rosati LM, Ng SK, Teboh Forbang R, Jackson J, Chang DT, Koong AC, Herman JM. Stereotactic body radiation therapy in pancreatic cancer: the new frontier. Expert Rev Anticancer Ther. 2014 Dec;14(12):1461-75. doi: 10.1586/14737140.2014.952286. Epub 2014 Sep 3. PMID 25183386
- [Background] Berber B, Sanabria JR, Braun K, Yao M, Ellis RJ, Kunos CA, Sohn J, Machtay M, Teh BS, Huang Z, Mayr NA, Lo SS. Emerging role of stereotactic body radiotherapy in the treatment of pancreatic cancer. Expert Rev Anticancer Ther. 2013 Apr;13(4):481-7. doi: 10.1586/era.13.19. PMID 23560842
- [Derived] Zhu X, Cao Y, Lu M, Zhao X, Jiang L, Ye Y, Ju X, Zhang H. Stereotactic body radiation therapy with sequential S-1 for patients with locally advanced pancreatic cancer and poor performance status: An open-label, single-arm, phase 2 trial. Radiother Oncol. 2021 Sep;162:178-184. doi: 10.1016/j.radonc.2021.07.009. Epub 2021 Jul 16. PMID 34274393
- [Derived] Zhu X, Ju X, Cao F, Fang F, Qing S, Shen Y, Jia Z, Cao Y, Zhang H. Safety and efficacy of stereotactic body radiation therapy combined with S-1 simultaneously followed by sequential S-1 as an initial treatment for locally advanced pancreatic cancer (SILAPANC) trial: study design and rationale of a phase II clinical trial. BMJ Open. 2016 Dec 1;6(12):e013220. doi: 10.1136/bmjopen-2016-013220. PMID 27909037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from February 2016 to March 2018 in Changhai Hospital affiliated to Navy Medical University.
Pre-assignment Details: There were significant events that occur after participant enrollment, but prior to assignment of participants to an arm or group.
Period: Overall Study
Arm/Group | Combination of Cyberknife With S-1
Started | 63
Completed | 53
Not Completed | 10
Not completed — disease progression | 10

BASELINE CHARACTERISTICS:
Population: Patients were enrolled according to the inclusion and exclusion criteria. All patients received follow-ups and were included in the final analysis.
Groups:
- Combination of Cyberknife With S-1: Patients with locally advanced pancreatic cancer meeting all inclusion criteria will receive combination of Cyberknife with S-1.
  combination of Cyberknife with sequential S-1: Radiation therapy combined with sequential chemotherapy
Arm/Group | Combination of Cyberknife With S-1
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 76.0 [71.5 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 63
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 63

OUTCOME MEASURES:

1. Primary Outcome: One-year Overall Survival Rate
Description: One-year overall survival rate is calculated by the ratio of number of patients surviving more than 1 year to the total number of patients enrolled.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Cyberknife With S-1
Number analyzed (Participants) | 63
Participants | 46

2. Secondary Outcome: Number of Participants With Acute Toxicities Following SBRT
Description: The acute toxicities are determined by RTOG Acute Radiation Morbidity Scoring Criteria.
Time Frame: Within 90 days after completion of SBRT
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Cyberknife With S-1
Number analyzed (Participants) | 63
Participants | 9

3. Secondary Outcome: Number of Participants With Late Toxicities Following SBRT
Description: The late toxicities are determined by RTOG/EORTC Late Radiation Morbidity Scoring Criteria.
Time Frame: 90 days after SBRT
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Cyberknife With S-1
Number analyzed (Participants) | 63
Participants | 5

4. Secondary Outcome: The Median Progression Free Survival Time Will be Determined.
Description: Progression-free survival is the time from the date of enrollment to the confirmation of disease progression at any sites, including local progression or metastasis, or death from any causes, if this occurred before disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination of Cyberknife With S-1
Number analyzed (Participants) | 63
months | 10.1 [9.7 to 10.5]

5. Secondary Outcome: The Quality of Life Will be Analyzed.
Description: The analysis of quality of life is based on The European Organization for Reasearch and Treatment of Cancer (EORTC): Quality of Life Questionnare-Core 30 (QLQ-C30). Higher scores in function domains and global health status indicate better quality of life, while higher scores in symptom domains imply worse quality of life. The scale range of all domains of QLQ-C30 is 0-100 (the minimum and maximum score is 0 and 100 points, respectively).
Time Frame: 1 years
Population: All domains of QLQ-C30 at 6 months after treatment are reported. Higher scores in function domains and global health status indicate better quality of life, while higher scores in symptom domains imply worse quality of life. The scale range of all following domains is 0-100 (the minimum and maximum score is 0 and 100 points, respectively).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Combination of Cyberknife With S-1
Number analyzed (Participants) | 63
units on a scale
  Global health status | 50.0 [33.3 to 66.7]
  Physical functioning | 64.2 [46.7 to 80.0]
  Role functioning | 54.8 [16.7 to 83.3]
  Emotional functioning | 68.5 [41.7 to 83.3]
  Cognitive functioning | 73.8 [33.3 to 83.3]
  Social functioning | 74.6 [33.3 to 83.3]
  Fatigue | 46.7 [33.3 to 66.7]
  Nausea and vomiting | 55.3 [33.3 to 83.3]
  Pain | 48.7 [33.3 to 83.3]
  Dyspnea | 9.5 [0 to 33.3]
  Insomnia | 19.0 [0 to 66.7]
  Appetite loss | 59.2 [33.3 to 100.0]
  Constipation | 13.2 [0 to 33.3]
  Diarrhea | 13.7 [0 to 33.3]
  Financial difficulties | 31.2 [0 to 66.7]

6. Secondary Outcome: Median Overall Survival Will be Determined.
Description: Median overall survival is calculated by Kaplan-Meier method.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination of Cyberknife With S-1
Number analyzed (Participants) | 63
months | 14.4 [13.2 to 15.6]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Radiation-induced acute toxicities are adverse effects that occur within 90 days after treatment, and determined by the Radiation Therapy Oncology Group, "Acute radiation morbidity scoring criteria". Late toxicities occurring three months after SBRT are evaluated by the Radiation Therapy Oncology Group/European Organization for Research on the Treatment of Cancer, "Late radiation morbidity scoring schema".
Arm/Group | Combination of Cyberknife With S-1
All-Cause Mortality (participants affected / at risk) | 63/63
Serious Adverse Events (participants affected / at risk) | 6/63
Other Adverse Events (participants affected / at risk) | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of Cyberknife With S-1 (N=63)
nausea and vomitting (Gastrointestinal disorders) | 6 (6) — Radiation-induced acute toxicities are adverse effects that occur within 90 days after treatment, and determined by the Radiation Therapy Oncology Group, "Acute radiation morbidity scoring criteria".

LIMITATIONS AND CAVEATS:
Lacks of comparison of gemcitabine alone or palliative radiotherapy recommended in NCCN guideline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT02704143/Prot_SAP_001.pdf